CLINICAL TRIAL: NCT07144397
Title: Does Concomitant Transobturator Lateral Suspension Improve Anterior Colporrhaphy Outcomes? A Randomized Controlled Trial
Brief Title: Transobturator Lateral Suspension in Anterior Colporrhaphy
Acronym: TLSAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Maribor (Other)
Responsible Party: Principal Investigator, Rok Sumak, Assistant, University Medical Centre Maribor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UKC-MB-KME-10/22
Record Dates: First submitted 2025-08-13; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Anterior Vaginal Wall Prolapse; Pelvic Organ Prolapse
Keywords: anterior colporrhaphy; transobturator lateral suspension; native tissue repair; randomized controlled trial; pelvic organ prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterior Colporrhaphy (AC) (No Intervention): Standard midline plication of pubocervical fascia using absorbable sutures under local anesthesia
- AC + Transobturator Lateral Suspension (TOLS) (Experimental): In addition to AC, bilateral non-absorbable sutures placed at the lateral edge of the pubocervical fascia, passed through obturator foramen, to provide lateral support
  Interventions: Procedure: TOLS

INTERVENTIONS:
Procedure: TOLS — "Standard AC plus bilateral lateral suspension using non-absorbable sutures passed through the obturator foramen to support lateral vaginal wall."
  Arms: AC + Transobturator Lateral Suspension (TOLS)

SUMMARY:
Anterior colporrhaphy (AC) is commonly used for anterior vaginal wall prolapse, but suffers high recurrence rates. This randomized trial assessed whether adding transobturator lateral suspension (TOLS) to AC decreases objective recurrence without compromising patient outcomes. In a cohort of 44 women (POP-Q ≥ 2), AC alone was compared to AC+TOLS over a 1-year follow-up. Results showed significantly lower objective recurrence with the added suspension.

DETAILED DESCRIPTION:
Conducted prospectively at University Medical Centre Maribor (Slovenia), this single-surgeon RCT randomized women with symptomatic anterior vaginal prolapse (POP-Q stage ≥ 2) to receive either standard AC or AC plus bilateral TOLS via non-absorbable suture across the obturator foramen. Primary outcome was objective anatomical recurrence (POP-Q ≥ 2) at 1 year. Secondary outcomes included subjective recurrence, satisfaction (Likert), operative time, postoperative and pelvic sidewall pain, and validated QOL instruments (UIQ-7, CRAIQ-7, POPIQ-7, PFIQ, POPDI-6, UDI-6, PFDI, PISQ).

ELIGIBILITY:
Inclusion Criteria:

* Adult women with symptomatic anterior vaginal wall prolapse (POP-Q stage ≥ 2)
* Eligible for native tissue repair
* Provided written informed consent

Exclusion Criteria:

* Previous anterior vaginal wall prolapse repair
* Predominant apical or posterior compartment defect

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-11-23 (Actual)

PRIMARY OUTCOMES:
Objective Recurrence Rate | 1 year postoperative
  Anatomical recurrence defined as POP-Q stage ≥ 2 in anterior compartment

SECONDARY OUTCOMES:
Subjective Recurrence Rate | 1 year postoperative
  Subjective recurrence was determined by a positive response to the validated question: "Do you usually have a bulge or something falling out that you can see or feel in your vaginal area?"
Patient Satisfaction | 1 year postoperative
  5-point Likert scale at 1 year
Operative time | 1 year postoperative
  Measured in minutes during surgery.
Postoperative Pain | 1 year postoperative.
  Assessed via VAS at discharge and immediate postoperative period
Pelvic Sidewall Pain | 1 year postoperative.
  Assessed at 1 year postoperative clinical examination, by pressing on obutrator membrane. Assesed as present or absent.

CONTACTS AND LOCATIONS:
Overall Officials: Rok Sumak, Principal Investigator — University Medical Centre Maribor, Department of General Gynaecology and Urogynaecology, Maribor, Slovenia
Locations (1):
- University Medical Centre Maribor, Maribor, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in this article, including baseline characteristics, intraoperative details, and outcome measures (objective recurrence, subjective recurrence, patient satisfaction, operative time, postoperative pain scores, and quality-of-life questionnaire scores), will be available to researchers upon reasonable request. Data will be shared beginning 6 months after publication of the main results and ending 5 years after article publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Start immediately, until 2027
Access Criteria: Access will be granted to investigators who provide a methodologically sound proposal, subject to approval by the corresponding author and the Institutional Ethics Committee. Data will be shared via a secure institutional repository following signing of a data access agreement.